CLINICAL TRIAL: NCT05455541
Title: Reliability of Artificial Intelligence (AI)-Augmented Point-of-care Cardiac Ultrasound (POCCUS) in the Hands of Internists
Brief Title: Reliability of Artificial Intelligence (AI)-Augmented Point-of-care Cardiac Ultrasound in the Hands of Internists
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: SHEBA-22-9419-KR-CTIL
Record Dates: First submitted 2022-07-03; First posted 2022-07-13 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-10

CONDITIONS: Cardiovascular Diseases; Valvular Heart Disease
MeSH Terms: conditions — Cardiovascular Diseases; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Hospitalized patients with an indication for POCUS examination: Patient with an accepted indication for point of care echo study that are clinical stable.
  Interventions: Diagnostic Test: AI augmented POCUS examination

INTERVENTIONS:
Diagnostic Test: AI augmented POCUS examination — Internists will perform POCUS studies as they consider appropriate for patient management. Interpretation of the POCUS exams will be aided by machine learning based analysis of the videos.

SUMMARY:
The study aim is to test the diagnostic performance of internists interpreting echo images aided by the AISAP CARDIO V0.7 diagnostic support system. Ground truth will be established by an interpretation by cardiologists specialized in echo, of the same POCUS images (acquired by the internist \ sonographer ).

Up to 1000 subjects; Study population will be distributed according to the following schema:

Group 1 -up to 800 patients hospitalized in the Internal Medicine division Group 2 - up to 200 patients hospitalized in the acute Geriatric division

ELIGIBILITY:
Inclusion Criteria:

1. Clinically indicated POCUS cardiac assessment as determined by the treating physicians for an accepted clinical indication
2. Willing and able to provide consent for a short partial transthoracic POCCUS examinations
3. No urgent or other compelling need for a comprehensive echo exam by the echo lab.

Exclusion Criteria:

1. Unstable clinical condition that does not permit any reasonable delay necessary to obtain consent and perform the POCCUS
2. Severe thoracic deformation or thoracic wall infection or wound that does not permit an adequate echocardiographic examination
3. Very poor or non-diagnostic echocardiographic imaging quality on prior echocardiography examinations.
4. Patients after lung resection
5. Patients unable lie in bed and undergo a standard echo study
6. Participation in an interventional study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospitalized patients in the internal medicine or geriatrics department that have an accepted indication for a POCUS study
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-08-21 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Degree of agreement | 30 days
  Agreement between the internists AI-aided interpretation and the interpretation by expert cardiologist
Clinical significant findings detected by the internist utilizing AI-aided POCUS | 30 days

SECONDARY OUTCOMES:
Percent of POCUS images of good quality | 30 days
Loops that AI interpreted | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fisher L, Fiman M, Segal E, Lidar S, Rubin N, Am-Shalom A, Cohen I, Faierstein K, Tsur AM, Schwammenthal E, Klempfner R, Zimlichman E, Raanani E, Maor E. Artificial intelligence assessment of valvular disease and ventricular function by a single echocardiography view. Front Digit Health. 2026 Jan 12;7:1684933. doi: 10.3389/fdgth.2025.1684933. eCollection 2025. PMID 41602208
- [Derived] Faierstein K, Fiman M, Loutati R, Rubin N, Manor U, Am-Shalom A, Cohen-Shelly M, Blank N, Lotan D, Zhao Q, Schwammenthal E, Klempfner R, Zimlichman E, Raanani E, Maor E. Artificial Intelligence Assessment of Biological Age From Transthoracic Echocardiography: Discrepancies with Chronologic Age Predict Significant Excess Mortality. J Am Soc Echocardiogr. 2024 Aug;37(8):725-735. doi: 10.1016/j.echo.2024.04.017. Epub 2024 May 11. PMID 38740271